CLINICAL TRIAL: NCT03713216
Title: Comparison of the Efficacy and Safety of NALDEBAIN With Conventional Treatment After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402
Record Dates: First submitted 2018-07-16; First posted 2018-10-19 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naldebain (Experimental): Subjects will receive one dose of Naldebain before surgery.
  Interventions: Drug: Naldebain
- Morphine (Active Comparator): Subjects will receive morphine after surgery.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Naldebain — 150 mg Nalbuphine sebacate
  Arms: Naldebain
Drug: Morphine — Morphine
  Arms: Morphine

SUMMARY:
To determine the effect and safety of NALDEBAIN versus Morphine as needed in patients after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This is an open-labeled, randomized clinical trial. Group A will receive one dose of NALDEBAIN before surgery. Group B will receive morphine as needed. Pain will be assessed for PACU, 4, 24, 48, 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with 20 years old or older.
2. Scheduled to electively undergo laparoscopic cholecystectomy.
3. Ability and willingness to provide informed consent.

Exclusion Criteria:

1. Not willing to adhere to the study visit schedule and complete all study assessments.
2. History of hypersensitivity or allergy to opioid, or NSAIDs or sesame oil.
3. Any clinically significant condition that may interfere with study assessments or compliance.
4. Pregnant or breastfeeding.
5. Medical history may cause abnormal intracranial pressure.
6. History of dependency, addiction, and withdrawal for narcotic drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | 24 hours after surgery
  Using visual analog scale (VAS) with grades from 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Consumption of supplemental analgesics | From Day 0 to Day 3
  Sum of supplemental analgesics

OTHER OUTCOMES:
Incidence of adverse event | From Day 0 to Day 3
  Times and incidence of adverse events (injection site reaction, vomiting, nausea, dizziness)
Percentage of Patient satisfaction | Day 3
  Percentage of patient satisfaction by 5-grade with 'highly satisfied', 'satisfied', 'uncertain', 'dissatisfied' or 'very dissatisfied'.

CONTACTS AND LOCATIONS:
Overall Officials: Sing-Ong Lee, MD, Principal Investigator — Cathay General Hospital
Locations (1):
- Cathay General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee SO, Huang LP, Wong CS. Preoperative Administration of Extended-Release Dinalbuphine Sebacate Compares with Morphine for Post-Laparoscopic Cholecystectomy Pain Management: A Randomized Study. J Pain Res. 2020 Sep 9;13:2247-2253. doi: 10.2147/JPR.S263315. eCollection 2020. PMID 32982387